CLINICAL TRIAL: NCT04374825
Title: Optimizing Quality of Life in Women Living With Metastatic Breast Cancer: Feasibility and Preliminary Efficacy of a Tailored, eHealth Supportive Oncology Intervention
Brief Title: Optimizing Quality of Life in Women Living With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Patricia Moreno, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SP0048722; STU00209333 (Other: Northwestern University Institutional Review Board); IRG-18-163-24 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic female breast cancer; Acceptance and Commitment Therapy; Stress management; eHealth
MeSH Terms: conditions — Breast Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Patients participating in the online pilot will be randomized to 1 of 3 study arms: 1) a usual care control, 2) CBSM, and 3) ACT. Women taking part in the intervention trial (i.e. women living with Stage IV [M1] breast cancer) will complete self-report psychosocial measures online at four assessments. Change across time will be assessed from baseline to mid-intervention (Week 4 of 8), immediately post-intervention (Week 8), and a one month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and Commitment Therapy (ACT) (Experimental): Weekly video conference groups led by a trained facilitator introducing key concepts of ACT
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Cognitive Behavioral Stress Management (CBSM) (Active Comparator): Weekly video conference groups led by a trained facilitator introducing key concepts of CBSM
  Interventions: Behavioral: Cognitive Behavioral Stress Management (CBSM)
- Usual care (No Intervention): Patients' usual health care as received over the duration of the pilot trial

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — This intervention consists of 8, 90-minute online group sessions delivered via video conference. Content will be developed by tailoring an ACT intervention to the specific needs of women with MBC, by using qualitative data gathered in patient focus groups. The intervention will incorporate key concepts of ACT (i.e., creating meaning and purpose in life via coping skills, activities in line with patients' values, and mindfulness meditation).
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Cognitive Behavioral Stress Management (CBSM) — This intervention consists of 8, 90-minute online group sessions delivered via videoconference. Content is drawn from a standard published CBSM intervention previously tested in other studies. The intervention incorporates key concepts of CBSM (i.e., managing stress via deep breathing and relaxation, identifying distorted thoughts,cognitive restructuring, and effective interpersonal communication).
  Arms: Cognitive Behavioral Stress Management (CBSM)

SUMMARY:
The purpose of this study is to develop and tailor an intervention program to improve the quality of life in women living with metastatic breast cancer. In the first phase of this study, we conducted patient focus groups to gather information about the unique challenges of living with MBC and what kinds of support women would like to receive in a tailored Acceptance and Commitment Therapy (ACT) intervention. In the second phase of the study, we will conduct a three-arm randomized controlled trial to the tailored ACT intervention with both a Cognitive Behavioral Stress Management (CBSM) intervention and usual care. The CBSM and ACT intervention groups will meet with a trained facilitator and 8-9 other patients, once per week via videoconference for 90 minute sessions over the course of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with metastatic (stage IV [M1]) female breast cancer, via physician diagnosis and confirmed through staff review of electronic medical record (i.e. imaging, surgical pathology reports, etc.).
* Patients must be comfortable speaking English for participation in group sessions.
* Patients must be age ≥ 18 years.
* Patients taking part in the 8 week online pilot trial must have a physician-anticipated life expectancy of > 6 months.
* Patients must have the ability to understand, and the willingness to sign, a written informed consent prior to registration on study.

Exclusion Criteria:

* Patients who have severe or impairing psychiatric illness/social situations that would limit compliance with study requirements are not eligible to enroll.
* Patients with early stage/non metastatic breast cancer (Stages I-III) are not eligible to enroll.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life (HRQoL) | Approx. 3 months
  Using the previously validated NIH PROMIS profile, change in HRQoL will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.
Change in wellbeing and disease symptom bother | Approx. 3 months
  Using the previously validated Functional Assessment of Cancer-Therapy-Breast (FACT-B), change in wellbeing and symptom bother will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.

SECONDARY OUTCOMES:
Change in meaning and purpose in life and positive affect | Approx. 3 months
  Using the previously validated PROMIS Short Forms for Meaning and Purpose and Positive Affect, change in meaning and purpose in life and positive affect will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.
Change in social support | Approx. 3 months
  Using the previously validated PROMIS Short Forms for Social Isolation, Emotional Support, and Informational Support, change in social support will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.

OTHER OUTCOMES:
Change in coping self-efficacy | Approx. 3 months
  Using the previously validated Measure of Current Status (MOCS) Self-Efficacy Scale, change in coping self-efficacy will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.
Change in acceptance | Approx. 3 months
  Using the previously validated Acceptance and Action Questionnaire-II, change in acceptance will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.
Change in open and engaged state | Approx. 3 months
  Using the previously validated Open and Engaged State Questionnaire, change in open and engaged state will be assessed from baseline to 1. mid-intervention (week 4), 2. immediately post-intervention (week 8), and a 3. one month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States